CLINICAL TRIAL: NCT01368302
Title: Attention Bias Modification Treatment (ABMT) for Patients With Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 949-2010
Record Dates: First submitted 2011-05-31; First posted 2011-06-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Attention Bias Modification Treatment (ABMT)
Keywords: attention bias modification treatment; cognitive bias modification; attention training; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Bias Modification (ABM) (Experimental): Attention training via repeated trials of a dot-probe task intended to normalize threat-related attention biases.
  Interventions: Behavioral: Attention Bias Modification Treatment (ABMT)
- Placebo (Placebo Comparator): Attention training via repeated trials of a dot-probe task not intended to change threat-related attention patterns.
  Interventions: Behavioral: Attention Bias Modification Treatment (ABMT)

INTERVENTIONS:
Behavioral: Attention Bias Modification Treatment (ABMT) — Attention training using a computerized spatial attention task (dot-probe) modified to alter threat-related attention patterns.

SUMMARY:
Patients with Post Traumatic Stress Disorder (PTSD) will be randomly assigned to either Attention Bias Modification Treatment (ABMT) designed to normalize threat-related attention biases or a placebo control condition not designed to change attention patterns. Outcome measures will be Post Traumatic Stress Disorder (PTSD), depression, and anxiety symptoms as measured by gold standard questionnaires and symptom counts derived from structured clinical interviews.

We expect to see significant Post Traumatic Stress Disorder symptom reduction in the Attention Bias Modification Treatment (ABMT) group relative to the placebo control group in which no symptomatic relief is expected.

ELIGIBILITY:
Inclusion Criteria:

* Combat-related PTSD diagnosis

Exclusion Criteria:

* Other treatment

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS) | 40 minutes
  The clinician-Administered PTSD Scale (CAPS) is a 30-item structured interview that corresponds to the DSM-IV criteria for PTSD (Blake, Weathers, Nagy, Kaloupek, Charney, & Keane, 1995).

SECONDARY OUTCOMES:
PTSD Check List (PCL) | 10 minutes
  Post-traumatic Stress symptoms will be evaluated using the 17-item National Center for PTSD Checklist of the Department of Veterans Affairs- PCL (Blanchard, Jones-Alexander, Buckley, & Forneris, 1996; Hoge, 2004; Kang, Natelson, Mahan, Lee, & Murphy, 2003).

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

REFERENCES:
- [Background] Hakamata Y, Lissek S, Bar-Haim Y, Britton JC, Fox NA, Leibenluft E, Ernst M, Pine DS. Attention bias modification treatment: a meta-analysis toward the establishment of novel treatment for anxiety. Biol Psychiatry. 2010 Dec 1;68(11):982-90. doi: 10.1016/j.biopsych.2010.07.021. PMID 20887977
- [Derived] Badura-Brack AS, Naim R, Ryan TJ, Levy O, Abend R, Khanna MM, McDermott TJ, Pine DS, Bar-Haim Y. Effect of Attention Training on Attention Bias Variability and PTSD Symptoms: Randomized Controlled Trials in Israeli and U.S. Combat Veterans. Am J Psychiatry. 2015 Dec;172(12):1233-41. doi: 10.1176/appi.ajp.2015.14121578. Epub 2015 Jul 24. PMID 26206075